CLINICAL TRIAL: NCT02307513
Title: A Phase 3, Multicenter, Randomized, Doubleblind, Placebo-controlled, Parallel Group Study, Followed by an Active-treatment Phase to Evaluate the Efficacy and Safety of Apremilast (CC-10004) in the Treatment of Subjects With Active Behcet's Disease
Brief Title: A Phase 3 Randomized, Double-blind Study to Evaluate the Efficacy and Safety of Apremilast (CC-10004) in Subjects With Active Behçet's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-10004-BCT-002; 2014-002108-25 (EudraCT Number)
Expanded Access: NCT03740516 (No longer available)
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Behçet's Syndrome
Keywords: APREMILAST (CC-10004); CC-10004; Efficacy; Safety; Phase 3; Behçet's Disease
MeSH Terms: conditions — Behcet Syndrome | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo / Apremilast (Experimental): Participants randomized to this arm will receive placebo tablets twice daily by mouth for the first twelve weeks followed by 52 weeks of 30 mg apremilast tablets twice daily by mouth.
  Interventions: Drug: Apremilast; Drug: Placebo
- Apremilast (Experimental): Participants randomized to this arm will receive 30 mg apremilast tablets twice daily by mouth for 64 weeks.
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Tablets for oral administration
  Other Names: Otezla®; CC-10004
Drug: Placebo — Tablets for oral administration
  Arms: Placebo / Apremilast

SUMMARY:
The main objective of this study is to evaluate the efficacy and safety of apremilast in the treatment of oral ulcers in adults with active Behçet's disease (BD).

DETAILED DESCRIPTION:
Behçet's disease, is a rare disorder that causes inflammation in blood vessels throughout the body. The signs and symptoms of Behçet's disease may include mouth sores, eye inflammation, skin rashes and lesions, and genital sores that vary from person to person and may come and go on their own. The exact cause of Behçet's is unknown, but it may be an autoimmune disorder, which means the body's immune system mistakenly attacks some of its own healthy cells.

This study will evaluate if apremilast is better than placebo (inactive substance in the same form as the drug) for the treatment of oral ulcers in subjects with active Behçet's disease. Other manifestations of the disease will also be assessed, such as, pain and tenderness in joints, eye inflammation, genital ulcers, and skin disease. This study also will test how well the body tolerates apremilast. In addition, the second purpose of the study is to assess the safety of apremilast in patients with Behçet's disease.

This study is a randomized, placebo-controlled, parallel design. The placebo-controlled period will be 12 weeks long and participants will receive apremilast or placebo. After the 12-week placebo-controlled period, all participants will receive apremilast for 52 weeks in the active treatment period. All participants will have their final study visit 4 weeks after stopping apremilast treatment.

Participants in Germany will have the opportunity to enter an optional open-label extension phase after the 52-week active treatment phase (week 64 visit), and continue until apremilast is commercially available for Behçet's disease or until apremilast is found not to be acceptable for Behçet's disease, according to either the sponsor or health authority.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures being conducted.
2. Male and female subjects ≥ 18 years of age at the time of signing the informed consent document.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Diagnosed with Behcet's disease meeting th4 International Study Group (ISG) criteria,
5. Oral ulcers that occurred at least 3 times in the previous 12-month period, including oral ulcers at the screening visit.
6. Subjects must have at least 2 oral ulcers at Visit 1 (Screening Visit), and:

   1. At least 2 oral ulcers at Visit 2 (day of randomization), when Visit 2 occurs at least 14 days after Visit 1. OR
   2. At least 3 oral ulcers at Visit 2 (day of randomization), when Visit 2 occurs at any time between 1 day and 42 days after Visit 1.
7. Have prior treatment with at least 1 non-biologic Behçet's disease therapy, such as, but not limited to, topical corticosteroids, or systemic treatment.
8. Candidate for systemic therapy, for the treatment of oral ulcers.

   a. A candidate for systemic therapy is a subject judged by the study Investigator as someone whose mucocutaneous ulcers are considered inappropriate for topical therapy based on the severity of disease and extent of the affected area, or whose oral ulcers cannot be adequately controlled by topical therapy.
9. Laboratory Measures: Must meet the following laboratory measures:

   * Hemoglobin > 9 g/dL
   * White blood cell (WBC) count ≥ 3000 /L(≥ 3.0 X 10^9/L) and ≤ 14,000/L (≤ 14 X 10^9/L )
   * Platelet count ≥ 100,000 /L (≥ 100 X 10^9/L)
   * Serum creatinine ≤ 1.5 mg/dL (≤ 132.6 μmol/L)
   * Total bilirubin ≤ 2.0 mg/dL
   * Aspartate transaminase (AST [serum glutamic oxaloacetic transaminase, SGOT]) and alanine transaminase (ALT [serum glutamate pyruvic transaminase, SGPT]) ≥ 1.5 X ULN. Subjects who fail screening due to ≥ 1.5 X ULN AST/SGOT and/or ALT/SGPT will be allowed to repeat AST/SGOT and/or ALT/SGPT tests within the screening phase. Repeat test results should be ≤ ULN (within reference range) to be eligible.

Laboratory tests will be allowed to be repeated 1 time if, in the Investigator's clinical judgment, there is a reasonable possibility of the repeat tests not meeting the exclusion values, and with concurrence from the Medical Monitor.

Contraception Requirements:

All Females of Child Bearing Potential (FCBP) must use one of the approved contraceptive options as described below while taking apremilast and for at least 28 days after administration of the last dose of the apremilast.

At the time of study entry, and at any time during the study when a FCBP's contraceptive measures or ability to become pregnant changes, the Investigator will educate the subject regarding contraception options and the correct and consistent use of effective contraceptive methods in order to successfully prevent pregnancy.

All FCBP must have a negative pregnancy test at Visits 1 and 2. All FCBP subjects who engage in activity in which conception is possible must use one of the approved contraceptive options described below:

Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; OR Option 2: Male or female condom (latex condom or non-latex condom NOT made out of natural [animal] membrane [for example, polyurethane]); PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.

Male subjects (including those who have had a vasectomy) who engage in activity in which conception is possible must use barrier contraception (latex or non-latex condoms NOT made out of natural [animal] membrane [for example, polyurethane]) while on IP and for at least 28 days after the last dose of IP.

Exclusion Criteria: The presence of any of the following will exclude a subject from the study enrollment.

Disease Specific Exclusions:

1. Behçet's disease-related active major organ involvement - pulmonary (eg, pulmonary artery aneurysm), vascular (eg, thrombophlebitis), gastrointestinal (eg, ulcers along the gastrointestinal tract), and central nervous systems (eg, meningoencephalitis) manifestations, and ocular lesions (eg, uveitis) requiring immunosuppressive therapy; however:

   1. Previous major organ involvement is allowed if it occurred at least 1 year prior to Visit 1 (Screening Visit) and is not active at time of enrollment.
   2. Subjects with mild BD-related ocular lesions not requiring systemic immunosuppressive therapy are allowed.
   3. Subjects with BD-related arthritis and BD-skin manifestations are also allowed.
2. Previous exposure to biologic therapies for the treatment of BD oral ulcers ( Previous biologic therapy exposure is allowed for other indications, including other manifestations of BD)
3. Prior use of apremilast.
4. Use of any investigational medication within 4 weeks prior to Visit 2 or 5 pharmacokinetic/pharmacodynamic half-lives (whichever is longer).
5. Current use of strong cytochrome P450 enzyme inducers (eg, rifampin, phenobarbital, carbamazepine, phenytoin)
6. Having received concomitant immune modulating therapy (except oral or topical corticosteroids) within:

   * Seven days prior to Visit 2 (Baseline Visit; day of randomization) for colchicines
   * Ten days prior to Visit 2 (Baseline Visit; day of randomization) for azathioprine and mycophenolate mofetil
   * Four weeks (28 days) prior to Visit 2 (Baseline Visit; day of randomization) for cyclosporine, methotrexate, cyclophosphamide, thalidomide, and dapsone.

   Note: Oral and topical corticosteroids must have been tapered as appropriate and discontinued prior to the day of Visit 2 (day of randomization).
   * At least 5 terminal half-lives for all biologics, including, but not limited to, those listed below; within:
   * Four weeks prior to Visit 2 (Baseline Visit; day of randomization) for etanercept
   * Eight weeks prior to Visit 2 (Baseline Visit; day of randomization) for infliximab
   * Ten weeks prior to Visit 2 (Baseline Visit; day of randomization) for adalimumab, golimumab, certolizumab, abatacept, and tocilizumab
   * Six months prior to Visit 2 (Baseline Visit; day of randomization) for secukinumab
7. Having received intra-articular or parenteral corticosteroids within 6 weeks (42 days) prior to Visit 2 (Baseline Visit; day of randomization).
8. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
9. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
10. Inability to provide voluntary consent.
11. Pregnant women or breast feeding mothers.
12. Systemic or opportunistic fungal infection.
13. Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections (including but not limited to tuberculosis and atypical mycobacterial disease, hepatitis B and C and herpes zoster, histoplasmosis, coccidiomycosis, but excluding onychomycosis) or any major episode of infection requiring hospitalization or treatment with IV or oral antibiotics within 4 weeks of the Screening Phase.
14. Clinically significant abnormality on chest radiograph.
15. Clinically significant abnormality on 12-lead electrocardiogram (ECG).
16. History of positive test for, or any clinical suspicion of, human immunodeficiency virus (HIV), or congenital or acquired immunodeficiency (eg, common variable immunodeficiency disease).
17. Malignancy or history of malignancy, except for:

    1. treated (ie, cured) basal cell or squamous cell in situ skin carcinomas;
    2. treated (ie, cured) cervical intraepithelial neoplasia (CIN) or carcinoma in situ of the cervix with no evidence of recurrence within the previous 5 years of Visit 1.
18. Any condition that confounds the ability to interpret data from the study.
19. Scheduled surgery or other interventions that would interrupt the subject's participation in the study.
20. Prior history of suicide attempt at any time in the subject's lifetime prior to Visit 2 (Baseline Visit; day of randomization) or major psychiatric illness requiring hospitalization within 3 years prior to Visit 2 (Baseline Visit; day of randomization).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2014-12-30 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2020-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (63):
- United States (11):
  - Arizona Arthritis and Rheumatology Research, PLLC, Phoenix, Arizona
  - University of California Davis Medical Center, Sacramento, California
  - Millennium Research, Ormond Beach, Florida
  - Arthritis and Rheumatology of Georgia, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Advanced Rheumatology, Lansing, Michigan
  - Shores Rheumatology, Saint Clair Shores, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - New York Methodist Hospital, Brooklyn, New York
  - NYU Langone Medical Center, New York, New York
  - University of Pennsylvania Health Systems, Philadelphia, Pennsylvania
- France (4):
  - Hopital de La Conception, Marseille
  - Pitié-Salpêtriere Hospital Paris, Paris
  - Hopital Cochin, Paris
  - Hospital Saint Louis, Paris
- Germany (3):
  - Charite Universitaetsmedizin Berlin, Berlin
  - Stadtisches Klinikum Dessau, Dessau
  - Asklepios Rheumazentrum Hamburg, Hamburg
- Greece (4):
  - Navy Hospital of Athens, Athens
  - Athens General Hospital 'G Gennimatas', Athens
  - Laiko General Hospital of Athens, Athens
  - Ippokratio General Hospital of Thessaloniki, Thessaloniki
- Israel (5):
  - Bnai Zion Medical Center, Haifa
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Organization, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
- Italy (3):
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Azienda Ospedaliera Regionale San Carlo, Potenza/Matera
  - Arcispedale Santa Maria Nuova, Reggio Emilia
- Japan (20):
  - Medical Hospital of Tokyo Medical and Dental University, Bunkyo-ku, Tokyo
  - Nippon Medical School Hospital, Bunkyō City
  - St. Luke's International Hospital, Chūōku
  - Tokyo Metropolitan Tama Medical Center, Fuchu-shi
  - Japanese Red Cross Society Himeji Hospital, Himeji-shi
  - Saitama Medical University Hospital, Iruma-gun, Saitama
  - Teikyo University Hospital, Itabashi-ku
  - Nihon University Itabashi Hospital, Itabashi-ku
  - St Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - University of Occupational and Environmentall Health, Kitakyushu
  - Kagawa University Hospital, Miki-cho
  - Saga Medical School Hospital, Saga
  - Kitasato University Hospital, Sagamihara
  - Sapporo Medical University Hospital, Sapporo, Hokkaidô
  - Hokkaido University Hospital, Sapporo, Hokkaidô
  - Shimonoseki City Hospital, Shimonoseki
  - Tokyo Medical University Hospital, Shinjyuku-ku
  - Tomishiro Central Hospital, Tomigusuku-shi
  - Ehime University Hospital, Tōon
  - Yokohama City University Hospital, Yokohama, Kanagawa
- Lebanon (3):
  - Hotel Dieu de France, Beirut
  - Ain Wazein Hospital, El Chouf
  - American University of Beirut Medical Center, El Chouf
- South Korea (5):
  - Chungnam National University Hospital, Daejeon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Konkuk University Hospital, Seoul
  - Ajou University Hospital, Suwon
- Turkey (Türkiye) (5):
  - Cukurova University Medical Faculty Balcali Hospital, Adana
  - Eskisehir Osmangazi University, Eskişehir
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Marmara University Hospital, Istanbul
  - Selcuk University Medical Faculty, Konya

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Mease PJ, Hatemi G, Paris M, Cheng S, Maes P, Zhang W, Shi R, Flower A, Picard H, Stein Gold L. Apremilast Long-Term Safety Up to 5 Years from 15 Pooled Randomized, Placebo-Controlled Studies of Psoriasis, Psoriatic Arthritis, and Behcet's Syndrome. Am J Clin Dermatol. 2023 Sep;24(5):809-820. doi: 10.1007/s40257-023-00783-7. Epub 2023 Jun 14. PMID 37316690
- [Derived] Hatemi G, Mahr A, Takeno M, Kim D, Melikoglu M, Cheng S, McCue S, Paris M, Chen M, Yazici Y. Impact of apremilast on quality of life in Behcet's syndrome: analysis of the phase 3 RELIEF study. RMD Open. 2022 Jul;8(2):e002235. doi: 10.1136/rmdopen-2022-002235. PMID 35798511
- [Derived] Hatemi G, Mahr A, Ishigatsubo Y, Song YW, Takeno M, Kim D, Melikoglu M, Cheng S, McCue S, Paris M, Chen M, Yazici Y. Trial of Apremilast for Oral Ulcers in Behcet's Syndrome. N Engl J Med. 2019 Nov 14;381(20):1918-1928. doi: 10.1056/NEJMoa1816594. PMID 31722152
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 53 sites in Europe (France, Germany, Greece, and Italy), Asia (Japan and the Republic of Korea), the United States, and Rest of the World (Israel, Lebanon, and Turkey).
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive either apremilast or placebo in a blinded fashion in the placebo-controlled treatment phase. After completion of 12 weeks, all participants were to receive apremilast for 52 weeks in the active treatment phase. Participants in Germany had the opportunity to enter an optional open-label extension phase at week 64.
  Participants were stratified by gender, history of uveitis and region (Japan and Other Regions).
Groups:
- Placebo/Apremilast: Participants received identically appearing placebo tablets twice a day (BID) from weeks 0 to 12 during the placebo-controlled treatment phase. At week 12 participants were switched to apremilast 30 mg tablets BID for 52 weeks during the active treatment phase and continued apremilast up to week 64.
  Participants in Germany had the option to continue receiving apremilast 30 mg BID in the extension phase.
- Apremilast: Participants received apremilast 30 mg tablets BID from weeks 0 to 12 during the placebo-controlled treatment phase and continued to receive apremilast 30 mg BID for 52 weeks during the active treatment phase up to week 64.
  Participants in Germany had the option to continue receiving apremilast 30 mg BID in the extension phase.
Period: Placebo Controlled Phase (Weeks 0-12)
Arm/Group | Placebo/Apremilast | Apremilast
Started | 103 | 104
Completed | 83 | 96
Not Completed | 20 | 8
Not completed — Adverse Event | 4 | 3
Not completed — Lack of Efficacy | 8 | 0
Not completed — Non-Compliance with Study Drug | 1 | 0
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 1
Period: Active Treatment Phase (Weeks 13-64)
Arm/Group | Placebo/Apremilast | Apremilast
Started | 83 | 95 (1 participant completed Week 12; did not enter into active treatment)
Completed | 68 | 75
Not Completed | 15 | 20
Not completed — Miscellaneous | 0 | 1
Not completed — Adverse Event | 4 | 9
Not completed — Lack of Efficacy | 2 | 2
Not completed — Withdrawal by Subject | 7 | 7
Not completed — Lost to Follow-up | 1 | 1
Not completed — Pregnancy | 1 | 0
Period: Long-term Extension
Arm/Group | Placebo/Apremilast | Apremilast
Started (Only participants in Germany had the option to continue receiving apremilast 30 mg BID in the extension phase.) | 2 | 0
Completed | 1 | 0
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: The intent to treat (ITT) population was defined as all randomized participants who received at least 1 dose of investigational product (IP). Participants were included in the treatment group to which they were originally randomized.
Groups:
- Placebo: Participants received identically appearing placebo tablets twice a day (BID) from weeks 0 to 12 during the placebo-controlled treatment phase. At week 12 participants were switched to apremilast 30 mg BID for 52 weeks during the active treatment phase and continued apremilast up to week 64.
- Apremilast 30 mg BID: Participants received apremilast 30 mg tablets BID from weeks 0 to 12 during the placebo-controlled treatment phase and continued to receive apremilast 30 mg BID for 52 weeks during the active treatment phase up to week 64.
- Total: Total of all reporting groups
Arm/Group | Placebo | Apremilast 30 mg BID | Total
Number analyzed (Participants) | 103 | 104 | 207
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.6 (12.66) | 39.4 (12.12) | 40.0 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 64 | 127
  Male | 40 | 40 | 80
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 30 | 32 | 62
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 1 | 1
  White | 68 | 69 | 137
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of the World [Count of Participants; unit: Participants]
  Europe | 27 | 25 | 52
  North America | 11 | 14 | 25
  Asia | 29 | 32 | 61
  Rest of World | 36 | 33 | 69
Duration of Behcet's Disease [Mean (Standard Deviation); unit: Years] — Population: One participant from each arm had duration of disease missing.
  Years
    number analyzed (Participants) | 102 | 103 | 205
    (all) | 6.94 (7.966) | 6.74 (7.397) | 6.84 (7.667)
Oral Ulcer Count [Mean (Standard Deviation); unit: Oral ulcers] | 3.9 (2.70) | 4.2 (3.65) | 4.1 (3.21)
Pain of Oral Ulcers Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: mm] — The oral ulcer pain visual analog scale ranges from 0 to 100 mm, with 0 mm representing no pain and 100 mm representing the worst possible pain. Population: Includes participants with available data.
  mm
    number analyzed (Participants) | 102 | 103 | 205
    (all) | 60.8 (26.92) | 61.2 (27.55) | 61.0 (27.17)
Behçet's Disease Current Activity Index (BDCAI) Score [Mean (Standard Deviation); unit: Units on a scale] — The BD Current Activity Index (as measured by the BD Current Activity Form) includes 12 questions regarding disease manifestations over the past 4 weeks, including oral and genital disease activity as well as manifestations involving the skin, joints, GI tract, eyes, nervous system, and vascular system. The BDCAI ranges from 0 to 12, where higher scores indicate a higher level of disease activity. Population: One participant from placebo arm had activity score index missing at baseline. Includes participants with available data.
  Units on a scale
    number analyzed (Participants) | 102 | 104 | 206
    (all) | 3.6 (1.67) | 3.7 (1.58) | 3.7 (1.62)
Behçet's Syndrome Activity Score (BSAS) [Mean (Standard Deviation); unit: scores on a scale] — The Behçet's Syndrome Activity Score contains 10 questions that assess the number of new oral and genital ulcers and skin lesions, gastrointestinal (GI), central nervous system (CNS), vascular, and ocular involvement, and the participant's current level of discomfort, each on a scale from 0 to 100 (worst). The item scores are totaled to create a score ranging from 0 to 100, with a higher score indicating a higher level of disease activity.
  scores on a scale | 44.30 (16.862) | 42.75 (16.224) | 43.52 (16.523)
Behçet's Disease Quality of Life (BD QoL) [Mean (Standard Deviation); unit: Units on a scale] — The BD QoL consists of 30 self-completed items that measure disease-related restrictions on the participant's activities and their emotional response to these restrictions. The BD QoL total score ranges from 0 to 30, with 0 representing no influence of BD on quality of life and 30 representing the greatest influence.
  Units on a scale | 11.24 (8.157) | 10.22 (8.245) | 10.73 (8.197)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) for the Number of Oral Ulcers From Baseline Through Week 12 (AUC W0-12)
Description: The number of oral ulcers that was counted for the analysis of the primary endpoint included current and recurrent ulcers at each time point; a single oral ulcer could be recounted multiple times if it persisted or recurred at subsequent visits.
Time Frame: Oral ulcers were assessed at weeks 0 (baseline), 1, 2, 4, 6, 8, 10, and 12 during the placebo-controlled period.
Population: The intent to treat (ITT) population included all randomized participants who received at least 1 dose of study drug. Multiple imputation (MI) was used to impute missing oral ulcer counts.
Measure: Least Squares Mean (Standard Error); unit: Ulcers*days
Groups:
- Placebo: Participants received identically appearing placebo tablets twice a day from weeks 0 to 12 during the placebo-controlled treatment phase.
- Apremilast 30 mg BID: Participants received apremilast 30 mg tablets BID from weeks 0 to 12 during the placebo-controlled treatment phase.
Arm/Group | Placebo | Apremilast 30 mg BID
Number analyzed (Participants) | 103 | 104
Ulcers*days | 222.14 (15.886) | 129.54 (15.943)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg BID; The AUC W0-12 for oral ulcer counts was compared between the placebo treatment group and the apremilast 30 BID treatment group using a 2-tailed parametric analysis of covariance (ANCOVA) test at the 0.05 significance level; Test type: Superiority; p < 0.0001, ANCOVA; ANCOVA model with AUC W0-12 as the response variables; treatment arm, sex, region as factors and the number of oral ulcers at baseline as a covariate; Difference in LS Mean = -92.60, 95% CI 2-sided [-130.59 to -54.60] — Treatment difference = Apremilast - Placebo

2. Secondary Outcome: Change From Baseline in Oral Ulcer Pain as Measured by Visual Analog Scale (VAS) at Week 12
Description: Pain of oral ulcers was measured using a 100 mm VAS scale. The participant was asked to draw a single line perpendicular to the VAS line at the point that represented the severity of their pain during the previous week, with 0 mm (the left-hand end of the scale) representing no pain and 100 mm (the right-hand end of the scale) representing the worst pain imaginable. The distance of the perpendicular line from the left-hand end of the scale was recorded.
  A negative change from baseline indicates improvement.
Time Frame: Baseline to week 12
Population: The ITT population with available baseline data. Last observation carried forward (LOCF) imputation was used. LOCF is the last observation (baseline value if no post-baseline assessment) is carried forward for missing values at week 12.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | Apremilast 30 mg BID
Number analyzed (Participants) | 102 | 103
mm | -15.9 (3.31) | -40.7 (3.34)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg BID; Test type: Superiority; p < 0.0001, ANCOVA; Based on an ANCOVA model for the change from baseline with the treatment arm, sex, region as factors and the baseline value as a covariate; Difference in LS Mean = -24.8, 95% CI 2-sided [-32.8 to -16.8]

3. Secondary Outcome: Change From Baseline in Disease Activity as Measured by Behçet's Syndrome Activity Score (BSAS) at Week 12
Description: The Behçet's Syndrome Activity Score (BSAS) contains 10 questions that assess the number of new oral and genital ulcers and skin lesions, GI, CNS, vascular, and ocular involvement, and the participant's current level of discomfort. The Behçet's Syndrome Activity Score ranges from 0 to 100, with a higher score indicating a higher level of disease activity. A negative change from baseline indicates improvement.
Time Frame: Baseline to week 12
Population: The intent to treat population with available baseline data. LOCF imputation was used for missing values at week 12.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Apremilast 30 mg BID
Number analyzed (Participants) | 103 | 104
Units on a scale | -5.41 (1.776) | -17.35 (1.796)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg BID; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Difference in LS Mean = -11.94, 95% CI 2-sided [-16.20 to -7.67]

4. Secondary Outcome: Change From Baseline in Disease Activity as Measured by Behçet's Disease Current Activity Form (BDCAF): Behçet's Disease Current Activity Index (BDCAI) at Week 12
Description: The Behçet's Disease Current Activity Form (BDCAF) consists of 3 component scores: the Behçet's Disease Current Activity Index (BDCAI) score, the Patient's Perception of Disease Activity, and the Clinician's Overall Perception of Disease Activity. The BDCAI consists of 12 questions regarding disease manifestations over the previous 4 weeks, including oral and genital disease activity, as well as other manifestations of BD involving the skin, joints, GI tract, eyes, nervous system, and vascular system. The BDCAI score is the sum score of 12 items and ranges from 0 to 12. A higher score indicates higher level of disease activity (worsening), and a negative change from baseline indicates improvement.
Time Frame: Baseline to week 12
Population: The intent to treat population with available baseline data. LOCF imputation was used for missing values at week 12.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Apremilast 30 mg BID
Number analyzed (Participants) | 102 | 104
Units on a scale | -0.4 (0.20) | -0.9 (0.20)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg BID; Test type: Superiority; p = 0.0335, ANCOVA; [statistical method as in outcome 2, analysis 1]; Difference in LS Means = -0.5, 95% CI 2-sided [-1.0 to -0.0]

5. Secondary Outcome: Change From Baseline in Disease Activity as Measured by Behçet's Disease Current Activity Form (BDCAF): Patient's Perception of Disease Activity at Week 12
Description: The Behçet's Disease Current Activity Form (BDCAF) consists of 3 component scores: the Behçet's Disease Current Activity Index (BDCAI) score, the Patient's Perception of Disease Activity, and the Clinician's Overall Perception of Disease Activity. The Patient's Perception of Disease Activity was assessed on a scale from 1 to 7, where a higher score indicates a higher level of disease activity and a negative change from baseline indicates improvement.
Time Frame: Baseline to week 12
Population: The intent to treat population with available data. LOCF imputation was used for missing values at week 12.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Apremilast 30 mg BID
Number analyzed (Participants) | 102 | 104
Units on a scale | -0.7 (0.18) | -1.7 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg BID; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Difference in LS Means = -1.0, 95% CI 2-sided [-1.4 to -0.6]

6. Secondary Outcome: Change From Baseline in Disease Activity as Measured by Behçet's Disease Current Activity Form (BDCAF): Clinician's Overall Perception of Disease Activity at Week 12
Description: The Behçet's Disease Current Activity Form (BDCAF) consists of 3 component scores: the Behçet's disease Current Activity Index (BDCAI) score, the Patient's Perception of Disease Activity, and the Clinician's Overall Perception of Disease Activity. The Clinician's Overall Perception of Disease Activity was assessed on a scale from 1 to 7, where a higher score indicates a higher level of disease activity and a negative change from baseline indicates improvement.
Time Frame: Baseline to week 12
Population: The intent to treat population with available baseline data. LOCF imputation was used for missing values at week 12.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Apremilast 30 mg BID
Number analyzed (Participants) | 102 | 104
Units on a scale | -0.7 (0.17) | -1.6 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg BID; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Difference in LS Means = -0.9, 95% CI 2-sided [-1.3 to -0.5]

7. Secondary Outcome: Percentage of Participants Who Achieved an Oral Ulcer Complete Response (Oral Ulcer-Free) by Week 6 and Remained Oral Ulcer-Free for at Least 6 Additional Weeks
Description: Participants who were oral ulcer-free by week 6 and remained oral ulcer-free for at least 6 consecutive weeks during the 12-week placebo-controlled treatment phase.
Time Frame: Baseline to week 12
Population: The intent to treat population
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Apremilast 30 mg BID
Number analyzed (Participants) | 103 | 104
Percentage of participants | 4.9 | 29.8
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg BID; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; 2 sided p-value based on the CMH test adjusting for sex and region; Adjusted difference in percentages = 25.1, 95% CI 2-sided [15.5 to 34.6] — Adjusted difference was the weighted average of the treatment differences across the 4 strata of combined sex and region factors with the CMH weights

8. Secondary Outcome: Time to Oral Ulcer Resolution (Complete Response)
Description: Time to oral ulcer resolution (defined as oral ulcer-free) was the time between the first dose date and the date when a complete response was achieved for the first time during the placebo-controlled treatment phase. For participants who did not achieve complete response or discontinued treatment before a complete response was achieved during the placebo-controlled treatment phase, time to event was censored at the last oral ulcer assessment date during the placebo-controlled treatment phase or the first dose date if there were no postbaseline ulcer assessments. Median and 95% confidence interval was based on Kaplan-Meier estimates.
Time Frame: Baseline to week 12
Population: The intent to treat population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Placebo | Apremilast 30 mg BID
Number analyzed (Participants) | 103 | 104
Weeks | 8.1 [4.7 to NA] — Could not be estimated due to the low number of events at the time of analysis | 2.1 [2.0 to 4.0]
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg BID; Test type: Superiority; p < 0.0001, Stratified Log-Rank Test; Treatment comparison is based on the stratified log-rank test, with sex and region as the stratification factors; Hazard Ratio (HR) = 2.400, 95% CI 2-sided [1.692 to 3.405] — The HR is based on the stratified Cox model with baseline number of oral ulcers and sex and region as the stratification factors

9. Secondary Outcome: Percentage of Participants Who Experienced an Oral Ulcer Complete Response at Week 12
Description: A complete response at week 12 was defined as participants who were oral ulcer free at week 12.
Time Frame: Week 12
Population: The intent to treat population; participants with missing data at week 12 were classified as non-responders.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Apremilast 30 mg BID
Number analyzed (Participants) | 103 | 104
Percentage of participants | 22.3 | 52.9
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg BID; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; 2 sided p-value based on the CMH test adjusting for sex and region; Adjusted difference in percentages = 30.6, 95% CI 2-sided [18.1 to 43.1] — [estimate comment as in outcome 7, analysis 1]

10. Secondary Outcome: Change From Baseline in Behçet's Disease Quality of Life (BD Qol) Scores at Week 12
Description: The Behçet's Disease Quality of Life questionnaire was developed to measure the influence of BD on a particpant's life. It consists of 30 self-completed itemized questions that measure disease-related restrictions on the participant's activities and their emotional response to these restrictions. The total score is the sum of all 30 items (each yes scores 1 and each no scores 0), with 0 representing no influence of Behçet's disease on a participant's quality of life and 30 representing the most severe influence. A negative change from baseline indicates improvement.
Time Frame: Baseline to week 12
Population: The intent to treat population. LOCF was used for missing values at week 12.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Apremilast 30 mg BID
Number analyzed (Participants) | 103 | 104
Units on a scale | -0.5 (0.66) | -3.5 (0.67)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg BID; Test type: Superiority; p = 0.0003, ANCOVA; [statistical method as in outcome 2, analysis 1]; Difference in LS Mean = -3.0, 95% CI 2-sided [-4.5 to -1.4]

11. Secondary Outcome: Percentage of Participants Who Experienced a Complete Response For Genital Ulcers at Week 12
Description: A genital ulcer complete response at week 12 was defined as participants who were genital ulcer-free at week 12.
Time Frame: Week 12
Population: The intent to treat population who had genital ulcers at baseline. Participants with missing data at week 12 were classified as non-responders.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Apremilast 30 mg BID
Number analyzed (Participants) | 17 | 17
Percentage of participants | 41.2 | 70.6
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg BID; Test type: Superiority; p = 0.1100, Cochran-Mantel-Haenszel; 2 sided p-value based on the CMH test adjusting for sex; Adjusted difference in percentages = 28.4, 95% CI 2-sided [-3.6 to 60.4] — Adjusted difference was the weighted average of the treatment differences across the 2 strata of sex with the CMH weights

12. Secondary Outcome: Percentage of Participants With no Oral Ulcers Following a Complete Response
Description: The definition includes participants who remained oral ulcer-free through week 12 after achieving a complete response (oral ulcer-free) prior to week 12.
Time Frame: Baseline to week 12
Population: The intent to treat population who had a complete response prior to week 12.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Apremilast 30 mg BID
Number analyzed (Participants) | 53 | 83
Percentage of participants | 13.2 | 31.3
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg BID; Test type: Superiority; p = 0.0204, Cochran-Mantel-Haenszel; Two-sided p-value was based on the CMH test, adjusting for sex and region; Adjusted difference in percentages = 17.5, 95% CI 2-sided [4.2 to 30.7] — [estimate comment as in outcome 7, analysis 1]

13. Secondary Outcome: Time to Recurrence of Oral Ulcers Following Loss of Complete Response
Description: Time to recurrence of oral ulcers following the loss of complete response (oral ulcer-free) was defined as the first instance when a participant had a reappearance of oral ulcers following a complete response, during the placebo-controlled treatment phase. For participants who did not have oral ulcer recurrence or discontinued treatment before any oral ulcer recurrence during the placebo-controlled treatment phase, time to event was censored at the last oral ulcer assessment during placebo-controlled treatment phase; For participants without any oral ulcer assessment following the first complete response, time to event was censored to the first complete response date.
Time Frame: Baseline through week 12
Population: The intent to treat population who had a complete response prior to week 12.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Placebo | Apremilast 30 mg BID
Number analyzed (Participants) | 53 | 83
Weeks | 2.3 [2.1 to 4.1] | 4.6 [3.1 to 6.1]
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg BID; Test type: Superiority; p = 0.0112, Stratified Log Rank Test; Treatment comparison is based on the stratified log-rank test, with sex and region as the stratification factors; Hazard Ratio (HR) = 0.611, 95% CI 2-sided [0.408 to 0.915] — [estimate comment as in outcome 8, analysis 1]

14. Secondary Outcome: Number of Oral Ulcers Following Loss of Complete Response Through Week 12
Description: Number of oral ulcers reported at the time of the first loss of complete response, ie, at the first instance when a participant had a reappearance of oral ulcers following a complete response, during the placebo-controlled treatment phase.
Time Frame: Baseline to week 12
Population: The intent to treat population who had a complete response prior to week 12.
Measure: Least Squares Mean (Standard Error); unit: oral ulcers
Arm/Group | Placebo | Apremilast 30 mg BID
Number analyzed (Participants) | 53 | 83
oral ulcers | 1.5 (0.21) | 1.1 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg BID; Test type: Superiority; p = 0.0683, ANCOVA; ANCOVA model with treatment group, sex and region as factors and the baseline ulcers number as a covariate; Difference in LS Means = -0.4, 95% CI 2-sided [-0.9 to 0.0]

15. Secondary Outcome: Change From Baseline in the Total Score of the Static Physician's Global Assessment (PGA) of Skin Lesions of BD at Week 12
Description: BD-related skin lesions (including acne-like lesions, folliculitis, and erythema nodosum) were evaluated according to the Static Physician's Global Assessment as follows:
  Score 0 = clear skin. Score 1 = mild in severity with the presence of 1 to 10 lesions (papules, pustules, cysts) or nodules at any anatomical site.
  Score 2 = Moderate severity; presence of 11 to 20 nodules or lesions (papules, pustules, cysts) at any anatomical site.
  Score 3 = Severe; presence of > 20 nodules or lesions (papules, pustules, cysts) at any anatomical site.
  The total sore was calculated as the sum of the acne-like lesions, folliculitis, and erythema nodosum scores, and therefore ranges from 0 to 9, where a higher score indicates a higher level of activity. A negative change from baseline indicates improvement.
Time Frame: Baseline to week 12
Population: The intent to treat population who had BD skin lesions at baseline. LOCF imputation was used for missing values at week 12.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Apremilast 30 mg BID
Number analyzed (Participants) | 59 | 58
scores on a scale | -0.8 (0.14) | -0.9 (0.14)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg BID; Test type: Superiority; p = 0.5944, ANCOVA; Based on an ANCOVA model for the change from baseline, with treatment arm, sex and region as factors and the baseline score as a covariate; Difference in LS Mean = -0.1, 95% CI 2-sided [-0.4 to 0.3]

16. Secondary Outcome: Change From Baseline in Genital Ulcer Pain as Measured by VAS Score at Week 12
Description: Pain of genital ulcers was measured using a 100 mm visual analog scale. The participant was asked to draw a single line perpendicular to the VAS line at the point that represented the severity of their pain during the previous week, with 0 mm (the left-hand end of the scale) representing no pain and 100 mm (the right-hand end of the scale) representing the worst pain imaginable. The distance of the perpendicular line from the left-hand end of the scale was recorded. A negative change from baseline indicates improvement.
Time Frame: Baseline to week 12
Population: The intent to treat population who had genital ulcers at baseline. The last observation (baseline value if no post-baseline assessment) was carried forward for missing values at week 12.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | Apremilast 30 mg BID
Number analyzed (Participants) | 17 | 17
mm | -24.5 (10.75) | -30.0 (11.22)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg BID; Test type: Superiority; p = 0.6182, ANCOVA; [statistical method as in outcome 15, analysis 1]; Difference in LS Mean = -5.5, 95% CI 2-sided [-27.6 to 16.7]

17. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) During the Placebo-controlled Treatment Period
Description: A TEAE is an adverse event (AE) with a start date on or after the date of the first dose of study drug and no later than 28 days after the last dose. An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. A serious AE (SAE) is any AE that resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect; or constituted an important medical event. For both AEs and SAEs the investigator assessed the severity of the event according to the grading scale:
  Mild: asymptomatic or with mild symptoms; Moderate: symptoms causing moderate discomfort and local or noninvasive intervention is indicated; Severe: symptoms causing severe discomfort or pain, symptoms requiring medical/surgical intervention.
Time Frame: From first dose of study drug in the placebo-controlled phase to the first dose of apremilast in the active treatment phase (12 weeks) or up to 28 days after last dose for participants who did not receive study drug at week 12, whichever was earlier.
Population: The safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Apremilast 30 mg BID
Number analyzed (Participants) | 103 | 104
Participants
  Any TEAE | 74 | 82
  Any Drug-related TEAE | 37 | 60
  Any Severe TEAE | 6 | 6
  Any Serious TEAE | 4 | 3
  Any TEAE Leading to Drug Interruption | 6 | 9
  Any TEAE Leading to Drug Withdrawal | 5 | 3
  Any TEAE Leading to Death | 0 | 0

18. Secondary Outcome: Number of Participants With TEAEs During the Apremilast-Exposure Period
Description: The apremilast-exposure period started on the date of the first dose of apremilast (week 0 for participants assigned to apremilast or week 12 for participants who were originally assigned to placebo and switched to apremilast at week 12) and ended 28 days after last dose in the active treatment phase.
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. An SAE is any AE that resulted in death; was life-threatening; required or prolonged inpatient hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect; or constituted an important medical event. The investigator assessed the severity of each event according to the grading scale:
  Mild: asymptomatic or mild symptoms; Moderate: symptoms causing moderate discomfort, local or noninvasive intervention indicated; Severe: symptoms causing severe discomfort or pain, requiring medical/surgical intervention.
Time Frame: From first dose of apremilast (week 0 for those assigned to apremilast or week 12 for those assigned to placebo) up to 28 days after last dose; up to 56 weeks and 68 weeks in each arm respectively.
Population: The apremilast as treated (AAT) population includes participants who received at least 1 dose of apremilast at any time during the study.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo/Apremilast: Participants received identically appearing placebo tablets BID from weeks 0 to 12 during the placebo-controlled treatment phase and switched to apremilast 30 mg BID tablets at week 12 and continued up through week 64.
- Apremilast/Apremilast: Participants received apremilast 30 mg tablets twice a day (BID) from weeks 0 to 12 during the placebo-controlled treatment phase and continued to receive apremilast 30 mg BID through week 64.
Arm/Group | Placebo/Apremilast | Apremilast/Apremilast
Number analyzed (Participants) | 83 | 104
Participants
  Any TEAE | 70 | 90
  Any Drug-related TEAE | 29 | 64
  Any Severe TEAE | 4 | 17
  Any Serious TEAE | 7 | 10
  Any TEAE Leading to Drug Interruption | 10 | 17
  Any TEAE Leading to Drug Withdrawal | 3 | 12
  Any TEAE Leading to Death | 0 | 0

ADVERSE EVENTS:
Time Frame: Placebo-controlled phase: From first dose of study drug to week 12 or up to 28 days after last dose for participants who did not receive study drug at week 12. Apremilast Exposure Phase: From first dose of apremilast (week 0 or week 12 for those assigned to placebo) up to 28 days after last dose; up to 56 weeks and 68 weeks in each arm respectively. Open-label extension: From first dose of apremilast in the extension phase to 28 days after last dose, up to 784 days.
Groups:
- Placebo-controlled Phase: Placebo: Participants received identically appearing placebo tablets twice a day from weeks 0 to 12 during the placebo-controlled treatment phase.
- Placebo-controlled Phase: Apremilast 30 mg BID: Participants received apremilast 30 mg tablets twice a day from weeks 0 to 12 during the placebo-controlled treatment phase.
- Apremilast Exposure Period: Apremilast 30 mg BID: Participants received apremilast 30 mg BID from week 0 or week 12 up to week 64.
- Open-label Extension Phase: Apremilast 30 mg BID: Participants in Germany received apremilast 30 mg BID in the open-label extension phase.
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg BID | Apremilast Exposure Period: Apremilast 30 mg BID | Open-label Extension Phase: Apremilast 30 mg BID
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/104 | 0/187 | 0/2
Serious Adverse Events (participants affected / at risk) | 4/103 | 3/104 | 17/187 | 0/2
Other Adverse Events (participants affected / at risk) | 52/103 | 67/104 | 132/187 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-controlled Phase: Placebo (N=103) | Placebo-controlled Phase: Apremilast 30 mg BID (N=104) | Apremilast Exposure Period: Apremilast 30 mg BID (N=187) | Open-label Extension Phase: Apremilast 30 mg BID (N=2)
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0 | 0
Genital infection (Infections and infestations) | 1 | 0 | 0 | 0
Genital infection fungal (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Infectious colitis (Infections and infestations) | 0 | 0 | 1 | 0
Lymph node tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 1 | 0
Vaginal stricture (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Arterial thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Behcet's syndrome (Vascular disorders) | 0 | 1 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-controlled Phase: Placebo (N=103) | Placebo-controlled Phase: Apremilast 30 mg BID (N=104) | Apremilast Exposure Period: Apremilast 30 mg BID (N=187) | Open-label Extension Phase: Apremilast 30 mg BID (N=2)
Dry eye (Eye disorders) | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 4 | 12 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 9 | 20 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 21 | 43 | 74 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 11 | 20 | 36 | 1
Vomiting (Gastrointestinal disorders) | 2 | 9 | 14 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 1
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 12 | 26 | 0
Urinary tract infection (Infections and infestations) | 4 | 1 | 2 | 1
Viral upper respiratory tract infection (Infections and infestations) | 5 | 7 | 20 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 6 | 18 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 8 | 16 | 0
Headache (Nervous system disorders) | 11 | 15 | 38 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 2
Insomnia (Psychiatric disorders) | 2 | 1 | 12 | 0
Behcet's syndrome (Vascular disorders) | 0 | 0 | 0 | 1
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is > 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 additional days. Investigator must delete confidential information before submission and defer publication to permit patent applications.

DOCUMENTS (2):
  • Study Protocol (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/13/NCT02307513/Prot_002.pdf
  • Statistical Analysis Plan (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/13/NCT02307513/SAP_000.pdf